CLINICAL TRIAL: NCT01821235
Title: A Single Centre, Single-blind, Randomized, Two-part, 6-way Cross-over Study to Investigate the Individual Bioequivalence of Gabasandoz® Relative to Neurontin® in Healthy Volunteers.
Brief Title: Evaluation of Individual Bioequivalence of Gabasandoz® Relative to Neurontin® in Healthy Volunteers
Acronym: DRUG13-GABA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EC/2013/210; 2013-001157-27 (EudraCT Number)
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Epilepsy and Neuropathic Pain
MeSH Terms: conditions — Epilepsy; Neuralgia | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Neurontin® (gabapentin) batch A (Experimental)
  Interventions: Drug: Neurontin® (gabapentin) batch A
- Neurontin® (gabapentin) batch B (Experimental)
  Interventions: Drug: Neurontin® (gabapentin) batch B
- Gabasandoz® (gabapentin) batch A (Experimental)
  Interventions: Drug: Gabasandoz® (gabapentin) batch A
- Gabasandoz® (gabapentin) batch B (Experimental)
  Interventions: Drug: Gabasandoz® (gabapentin) batch B

INTERVENTIONS:
Drug: Neurontin® (gabapentin) batch A — Neurontin® 800 mg tablets (gabapentin) batch A, given 2 times
  Arms: Neurontin® (gabapentin) batch A
Drug: Neurontin® (gabapentin) batch B — Neurontin® 800 mg tablets (gabapentin) batch B, given 1 time
  Arms: Neurontin® (gabapentin) batch B
Drug: Gabasandoz® (gabapentin) batch A — Gabasandoz® 800 mg tablets (gabapentin) batch A, given 2 times
  Arms: Gabasandoz® (gabapentin) batch A
Drug: Gabasandoz® (gabapentin) batch B — Gabasandoz® 800 mg tablets (gabapentin) batch A, given 1 time
  Arms: Gabasandoz® (gabapentin) batch B

SUMMARY:
The NO SWITCH list is based on the hypothesis that the pharmacokinetic differences between different batches of one medicines are smaller than the pharmacokinetic differences between two medicines (from a different manufacturer, e.g. brand versus generic medicine). The aim of this study is to investigate the hypothesis using gabapentin as test product. Therefore, the first objective of this study is to investigate the individual bioequivalence - or switchability - of Gabasandoz® 800 mg relative to Neurontin 800 mg®. The second objective is to investigate the individual bioequivalence between two different batches of the same medicine, for Gabasandoz® 800 mg and Neurontin® 800 mg.

DETAILED DESCRIPTION:
At the end of 2011, the Belgian Federal Agency for Medicines and Health Products (FAMHP) introduced a list of medicines, called the 'NO SWITCH' list1. This list contains 42 active pharmaceutical ingredients with a narrow therapeutic index (i.e. small differences between the effective and toxic concentration), very toxic ingredients and all antiepileptics. For the active ingredients on the NO SWITCH-list, the FAMHP advises, once treatment is started with a medicines from a particular manufacturer, to continue treatment with exactly the same medicine (from the same manufacturer). In other words, switching from e.g. Neurontin® 800 mg to Gabasandoz® 800 mg during treatment is not recommended. However, switching is possible, but only when done carefully and under the supervision of a physician.

The NO SWITCH list is based on the hypothesis that the pharmacokinetic differences between different batches of one medicines are smaller than the pharmacokinetic differences between two medicines (from a different manufacturer, e.g. brand versus generic medicine).

The aim of this study is to investigate the hypothesis using gabapentin as test product. Therefore, the first objective of this study is to investigate the individual bioequivalence - or switchability - of Gabasandoz® 800 mg relative to Neurontin 800 mg®. The second objective is to investigate the individual bioequivalence between two different batches of the same medicine, for Gabasandoz® 800 mg and Neurontin® 800 mg.

This is a two-parted study. The first part is a 6 way crossover pilot study with 12 healthy volunteers (men and women). Data from this pilot study will be used to determine the following pharmacokinetic parameters: AUC0-t, AUC, Cmax and T1/2. The obtained data will be used to develop a Limited Sampling Strategy (LSS), i.e. a strategy to determine AUC and Cmax from a limited number of plasma concentrations. A simulation study will be performed, using data from the pilot study to determine the amount of volunteers needed to result into an appropriate statistical power. This simulation study will be performed according to the FDA Guidance for Industry: Statistical Approaches to Establishing Bioequivalence2.

Part two of the study will be a 6 way crossover and AUC and Cmax will be determined using the developed Limited Sampled Strategy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged between 18 and 55 years at screening, extremes included.
* A Body Mass Index of 18.0 to 30.0 kg/m².
* Good physical and mental health.
* Subject is a non-smoker for at least 3 months prior to dosing.

Exclusion Criteria:

* Clinically relevant abnormal laboratory, ECG recordings, vital signs or physical findings at screening as judged by the investigator.
* History of hypersensitivity or idiosyncrasy to gabapentin or any other anti-convulsive agents.
* Positive serology for hepatitis B antigen, hepatitis C antibodies, HIV 1 or HIV 2 antibodies.
* History of alcohol or drug abuse within the last 2 years.
* Blood donation within 1 month before screening.
* Female subjects who are pregnant or lactating.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) and Peak Plasma Concentration (Cmax) of Neurontin® 800 mg | As of from dosing till 36 h postdose
  16 bloodsamples will be taken; Blood samples taken at 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 4.5h, 5h, 6h, 7h, 8h, 10h, 12h, 24h, 36h post-dose.
Area under the plasma concentration versus time curve (AUC) and Peak Plasma Concentration (Cmax) of Gabasandoz® 800 mg | As of from dosing till 36 h postdose
  16 bloodsamples will be taken; Blood samples taken at 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 4.5h, 5h, 6h, 7h, 8h, 10h, 12h, 24h, 36h post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Van Bortel, Phd, MD, Principal Investigator — UZ Ghent
Locations (1):
- Drug Research Unit Ghent (D.R.U.G.), Ghent, Belgium